CLINICAL TRIAL: NCT02841826
Title: Evaluation of a Novel and Simplified Technique for Intrauterine Contraceptive Devices Insertion: a Prospective Cohort Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIUD
Record Dates: First submitted 2016-07-20; First posted 2016-07-22 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I: IUD without uterine sound group (Other): Transvaginal ultrasound before to intrauterine contraceptive device insertion without uterine sounding.
  Interventions: Other: IUD; Radiation: Transvaginal ultrasound
- Group II: IUD with uterine sound (Other): Intrauterine contraceptive device inserted by classic method
  Interventions: Other: IUD; Other: Uterine sounding

INTERVENTIONS:
Other: IUD
Other: Uterine sounding
  Arms: Group II: IUD with uterine sound
Radiation: Transvaginal ultrasound
  Arms: Group I: IUD without uterine sound group

SUMMARY:
The intrauterine devices (IUDs) are a safe, reliable, long-acting and reversible contraceptive method. It is also sound safe and cheap contraceptive methods available and is nearly maintenance free for up to 10 years.

The fear and the pain associated with IUDs insertion consider barriers to using this contraception method, this is because that the mucosal lining of female genital tract is highly sensitive to touch and pain. However; most of small procedures done in this sensitive area are performed without analgesia.

The pain during IUDs insertion is due to application of the tenaculum , traction of the cervical canal, passing the uterine sound, insertion of the IUDs through the cervix, and irritation of the endometrial lining by the IUDs.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting intrauterine contraceptive device as a contraction
* Women accepted participation in the study

Exclusion Criteria:

* Uterine abnormalities
* Endometrial lesions as polyp
* Adenomyosis
* Fibroids distorting the cavity
* Intrauterine adhesions.
* Chronic pelvic pain
* Dysmenorrhea
* History of cervical surgery

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The degree of pain perception measured visual analogue score | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes